CLINICAL TRIAL: NCT04560894
Title: SCT-I10A in Combination With SCT510 Versus Sorafenib as First-Line Therapy for Advanced Hepatocellular Carcinoma (HCC): A Multicenter, Randomized, Open-label,Phase 2/3 Trial
Brief Title: SCT-I10A Plus SCT510 Versus Sorafenib as First-Line Therapy for Advanced Hepatocellular Carcinoma
Acronym: HCC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCT-I10A-C301
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCT-I10A+SCT510 (Experimental)
  Interventions: Drug: SCT-I10A; Drug: SCT510
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib 200mg

INTERVENTIONS:
Drug: SCT-I10A — Participants receive SCT-I10A intravenously，200mg，d1，Q3w
  Arms: SCT-I10A+SCT510
Drug: SCT510 — Participants receive SCT510 intravenously，15mg/kg，d1，Q3w
  Arms: SCT-I10A+SCT510
Drug: Sorafenib 200mg — Participants receive sorafenib orally，400mg bid
  Arms: Sorafenib

SUMMARY:
The purpose of the study is to assess the safety and effectiveness of SCT-I10A in combination with SCT510 in patients with HCC who have not received prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of HCC not suitable for radical surgery and/or local treatment，or progressed after surgery and/or local treatment.
* No prior systemic therapy for HCC(End of postoperative adjuvant chemotherapy for more than 6 months allowed).
* Child-Pugh ≤7 , no history of hepatic encephalopathy.
* Barcelona Clinic Liver Cancer stage B, not suitable for local treatment and BCLC C.
* At least one measurable lesion based on Recist1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Adequate hematologic and organ function.

Exclusion Criteria:

* Local treatment or surgery for liver lesions within 4 weeks.
* Prior liver or other organ transplantation.
* Active Central nervous system (CNS) metastasis or leptomeningeal metastases.
* Gastrointestinal perforation and/or fistula or intraperitoneal abscess within 6 months prior to the start of study treatment.
* Hemorrhage tendency or high-risk for bleeding , severe coagulation disorders.
* Active known, or suspected autoimmune disease.
* Any condition that is not suitable for participate in this study as determined by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 3years
Progression-free survival(PFS)evaluated by the Blinded Independent Central Review Committee (BICR) based on RECIST V1.1 | up to 3years

SECONDARY OUTCOMES:
PFS | up to 3years
  PFS evaluated by investigator based on RECIST V1.1
PFS | up to 3years
  PFS evaluated by BICR based on mRECIST.
Objective response rate (ORR) | up to 3years
  ORR evaluated by BICR based on RECIST V1.1.
ORR | up to 3years
  ORR evaluated by BICR based on mRECIST.
ORR | up to 3years
  ORR evaluated by investigator based on RECIST V1.1
Serum concentration of SCT-I10A and SCT510 | up to 3years
Anti-drug antibody (ADA) | up to 3years

CONTACTS AND LOCATIONS:
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhao C, Zhang Y, Wang G, Zheng J, Chen W, Lu Z, Zhuang L, Gu S, Han L, Zheng Z, Yu Z, Yang Y, Sun H, Wei X, Cheng Y, Lin H, Zhu B, Wu G, Lei K, Wang W, Wang Y, Chen K, Xu X, Zheng C, Bi Y, Ding S, Zhang J, Li W, Liu H, Wang J, Liu X, Du Y, Cai L, Wang J, Luo Z, Xing B, Shen J, Yang L, Wu J, Jiang O, Peng Z, Liu X, Cao B, Shen L, Xu A, Li A, Chen S, Fu T, Chen J, Jin C, Zhang L, Lv J, Zhang C, Zhang X, Wang Y, Su H, Zhou Q, Gai W, Xie L, Xu J. Finotonlimab (PD-1 inhibitor) plus bevacizumab (bevacizumab biosimilar) as first-tier therapy for late-stage hepatocellular carcinoma: a randomized phase 2/3 trial. Signal Transduct Target Ther. 2025 Aug 6;10(1):249. doi: 10.1038/s41392-025-02333-5. PMID 40769977